CLINICAL TRIAL: NCT05323669
Title: Study of Molecular-genetic Profile of Thyroid Nodules
Brief Title: Molecular Profile of Thyroid Nodules
Acronym: MPTN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Belarusian State Medical University (Other)
Collaborators: The Institute of Genetics and Cytology National Academy of Sciences of Belarus (Unknown); Minsk City Clinical Oncologic Centre (Unknown)
Responsible Party: Principal Investigator, Siarhei Yakubouski, MD PhD Assistant Professor, Belarusian State Medical University
Other Study IDs: 20220367
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Thyroid Cancer; Thyroid Nodule
Keywords: thyroid cancer; thyroid nodule; miRNA; molecular testing
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule | interventions — Molecular Diagnostic Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — histological samples (Formalin Fixed Paraffin Embedded tumour tissue (FFPE)) fixed cytological samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Molecular testing — Molecular testing of thyroid nodules

SUMMARY:
Profiling and comparative analysis of genomic alterations and miRNA expression in benign and malignant thyroid tumors using histological and cytological specimens will be performed. Obtained information is necessary to create a molecular test to refine the cancer risk of cytologically indeterminate thyroid nodules.

DETAILED DESCRIPTION:
This is an non-randomised retrospective study consisting of 2 parts. Part A. Histological specimens (formalin fixed paraffin embedded) of patients who were operated on for benign and malignant thyroid disorders will undergo molecular testing to create a molecular profile of thyroid nodules characteristic of Belarusian population.

Part B. Fixed cytological smears of indeterminate thyroid nodules (categories III, IV and V according to Bethesda scoring system) of operated patients will undergo molecular testing to evaluate the possibility and reliability of molecular testing of fixed cytological smears using available assays.

ELIGIBILITY:
Inclusion Criteria:

Patients operated on for malignant and benign thyroid tumors. Age is greater than or equal to 18 years old.

Exclusion Criteria:

no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of the Republic of Belarus
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-04-11 (Estimated); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular profile of thyroid nodules | 2 years
  To develop a molecular profile of thyroid nodules that will allow to distinguish benign from malignant tumor

CONTACTS AND LOCATIONS:
Overall Officials: Gennadij G Kondratenko, MD PhD Prof, Study Director — Belarusian State Medical University

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after summary data are published
Access Criteria: IPD will be shared through publications